CLINICAL TRIAL: NCT03653013
Title: Neuropsychological Consultation as Part of Pediatric Diabetes Care: Does it Improve Glycemic Control and Family Functioning?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-00649
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Diabetes; Glycinemia
MeSH Terms: conditions — Diabetes Mellitus | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Usual standard of care from their diabetes care team
  Interventions: Behavioral: Usual standard of care
- Neuropsychological Consultation Group (Experimental): Children will be administered a number of neuropsychological tests. Children and parents in Group 2 will also complete a pediatric quality of life scale (PedsQL, Generic Scale and Diabetes Module), diabetes related family conflict scale (DFCS-R) to assess quality of life and family stress at the start of the study, as well as the self-report form of the BRIEF-2 if they are over age 11. Parents will also undergo a brief literacy and numeracy screening using the Wide Range Achievement Test, complete a parent report assessing their children's executive functioning skills at the start of the study (BRIEF-2) and they will fill out the Family Impact Module.
  Interventions: Behavioral: Neuropsychological Consultation

INTERVENTIONS:
Behavioral: Usual standard of care — Participants will receive treatment and diabetes management as usual standard of care from their diabetes care team. They will also complete as part of the study visit: a pediatric quality of life scale(PedsQL,GenericScale and Diabetes Module) and diabetes related family conflict scale (DFCS-R) to assess quality of life and family stress at the start of the study.
  Other Names: Control Group
  Arms: Control Group
Behavioral: Neuropsychological Consultation — Children and parents in Group 2 will also complete a pediatric quality of life scale (PedsQL,Generic Scale and Diabetes Module),diabetes related family conflict scale (DFCS-R) to assess quality of life and family stress at the start of the study, as well as the self-report form of the BRIEF-2 if they are over age 11. Parents will also undergo a brief literacy and numeracy screening using the Wide Range Achievement Test, complete a parent report assessing their children's executive functioning skills at the start of the study (BRIEF-2) and they will fill out the Family Impact Module.
  Arms: Neuropsychological Consultation Group

SUMMARY:
This is a randomized controlled open label study design (study team will not be blinded) to measure whether including targeted neuropsychological consultations as part of pediatric diabetes care informs treatment and educational planning, improves glycemic control, and improves quality of life. Patients will be randomized 1:1 ratio to Group 1-Control group and Group 2-Neuropsychological consultation group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with type 1 diabetes and followed for their care at the NYU pediatric diabetes center
* English speaking families

Exclusion Criteria:

* not english speaking
* diagnosed with type 1 diabetes within the last 6 months

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Improved Glycemic Control measured by assessment of glycemic control (HgbA1C) | 0 Months
Improved Glycemic Control measured by assessment of glycemic control (HgbA1C) | 3 Months
Improved Glycemic Control measured by assessment of glycemic control (HgbA1C) | 6 Months
Improved Glycemic Control measured by assessment of glycemic control (HgbA1C) | 9 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Gallagher, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.